CLINICAL TRIAL: NCT02831725
Title: An Observational Cohort Study to Establish Accurate Nutrition Therapy for Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-991
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Nutrition Therapy for Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
1. Demographics data;
2. Nutritional evaluation data;
3. All biochemical monitoring data during the study period;
4. All nutritional treatment data will be recorded daily during the study period, including actual calorie intake, protein intake, and the proportion of calorie/protein administered by EN and/or PN route. The nutritional treatment protocol will be decided by the attending physician, the investigator will not intervene.
5. A blood sample (5 ml) will be drawn from every patient immediately after they enroll into the study, and the metabolomics of the samples will be analyzed analysis using a combined 800 MHz 1H-NMR-UPLC-MS system. The data will then be used to establish metabolic profile baseline.
6. We will establish a sub-group that contains 20 patients (chosen from enrolled patients according to APACHE II scores: 10 patients are APACHE II scores in 21-30). We will take one blood sample daily during the whole study period. The plasma sample will be used for metabolomics analysis using an 800 MHz 1H-NMR-UPLC-MS system. And the data will be used for metabolic dynamic modeling.
7. Clinical outcomes data, which include: 1) Complications after the operation (intestinal fistula, pancreatic fistula, biliary fistula and sepsis, bleeding, nosocomial infection); 2) death event; 3) ICU-stay; 4) Length of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* age: 18-70
* patients are underwent Whipple operation or subtotal gastrectomy and ever admitted to intensive care unit (ICU) after the operation
* receive parenteral or enteral nutrition > 3 days

Exclusion Criteria:

* has metabolic disorders: diabetes, thyroid disease
* Pregnant or breastfeeding
* The presence of drug or alcohol dependence
* The presence of tuberculosis, HIV infection and other acute infectious disease
* Serious liver, kidney, heart and other vital organ failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized adult patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
complications after the operation | three years
  intestinal fistula, pancreatic fistula, biliary fistula and sepsis, bleeding, nosocomial infection